CLINICAL TRIAL: NCT00863889
Title: Steroid Injection for the Treatment of Greater Trochanteric Pain Syndrome: A Randomized Controlled Trial
Brief Title: Steroid Injection for the Treatment of Greater Trochanteric Pain Syndrome
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Thomas L Bradbury, MD, Residency Program Director, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00010776
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Last update posted 2013-09-23 (Estimated); Status verified 2013-09

CONDITIONS: Bursitis
MeSH Terms: conditions — Bursitis | interventions — Lidocaine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 1cc Depomedrol, 4 cc 1% Lidocaine, 4 cc 0.25% Marcaine
  Interventions: Drug: Depomedrol injection
- 2 (Placebo Comparator): 4 cc 1% Lidocaine, 4 cc 0.25% Marcaine
  Interventions: Drug: Lidocaine, Marcaine

INTERVENTIONS:
Drug: Depomedrol injection — 1 cc of Depomedrol 80
  Arms: 1
Drug: Lidocaine, Marcaine — 4 cc of each local anesthetic
  Arms: 2

SUMMARY:
The objective of this study is to conduct a randomized, single-blinded placebo controlled trial comparing two modalities for the treatment of pain and mobility associated with trochanteric bursitis: (1) injection of glucocorticosteroid and local anesthetic, (2) injection of local anesthetic. We hope to determine whether steroid injections provide a statistically significant improvement in pain symptoms and hip mobility in subjects with trochanteric bursitis, as compared to an injection of local anesthetic. Our null hypothesis is that no statistically significant difference exists between the two treatment modalities.

DETAILED DESCRIPTION:
Trochanteric bursitis is an inflammation of the bursal sac overlying the greater trochanter of the femur. The etiology of this disease is unknown, but it is clinically characterized by chronic aching pain over the lateral aspect of the hip, which can be exacerbated by certain movements such as external rotation and abduction (2). In order to objectively determine the level of pain and mobility associated with trochanteric bursitis, some orthopaedic surgeons use scoring systems (a qualitative and quantitative scoring test) to assess patients (4).

In our practice, trochanteric bursitis has been treated by injection of glucocorticosteroids (steroids) combined with local anesthetic at the site of the greater trochanter (1). Additionally, it has been found that increasing steroid dosage provides a greater level of relief (3). Although steroids are usually an effective treatment, no studies to date have compared steroid injections for relief of trochanteric bursitis pain and mobility versus a placebo injection or local anesthetic injection alone.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with tenderness at the greater trochanter

Exclusion Criteria:

* Subjects < 17 years of age
* Subjects with previous surgery to the greater trochanter
* Subjects allergic to Lidocaine, Marcaine, or Depomedrol

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-03; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
WOMAC hip score | 2 weeks, 6 weeks, 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Tom Bradbury, MD, Principal Investigator — Emory University
Locations (1):
- Dr. Tom Bradbury, Atlanta, Georgia, United States

REFERENCES:
- [Background] Shbeeb MI, O'Duffy JD, Michet CJ Jr, O'Fallon WM, Matteson EL. Evaluation of glucocorticosteroid injection for the treatment of trochanteric bursitis. J Rheumatol. 1996 Dec;23(12):2104-6. PMID 8970048
- [Background] Silva F, Adams T, Feinstein J, Arroyo RA. Trochanteric bursitis: refuting the myth of inflammation. J Clin Rheumatol. 2008 Apr;14(2):82-6. doi: 10.1097/RHU.0b013e31816b4471. PMID 18391676
- [Background] Brinks A, van Rijn RM, Bohnen AM, Slee GL, Verhaar JA, Koes BW, Bierma-Zeinstra SM. Effect of corticosteroid injection for trochanter pain syndrome: design of a randomised clinical trial in general practice. BMC Musculoskelet Disord. 2007 Sep 19;8:95. doi: 10.1186/1471-2474-8-95. PMID 17880718
- [Background] Baker CL Jr, Massie RV, Hurt WG, Savory CG. Arthroscopic bursectomy for recalcitrant trochanteric bursitis. Arthroscopy. 2007 Aug;23(8):827-32. doi: 10.1016/j.arthro.2007.02.015. Epub 2007 Jun 14. PMID 17681203